CLINICAL TRIAL: NCT00684619
Title: Phase II-Study With Nelarabine in Patients With Refractory Oder Relapsed T- ALL or T-lymphoblastic Lymphoma (Amend.7)
Brief Title: 506U78 In Relapsed Or Refractory Acute Lymphoblastic Leukemia (T-ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, GMALL Head, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LN_GMALLE_2004_55
Record Dates: First submitted 2008-05-16; First posted 2008-05-26 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: T-ALL, T-NHL (Lymphoblastic)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Nelarabine
  Interventions: Drug: Nelarabine

INTERVENTIONS:
Drug: Nelarabine — 1500 mg/m² i.v., duration 2 hrs, day 1, 3, 5
  Other Names: Compound 506U78; Atriance; Arranon

SUMMARY:
The purpose of this study is to determine whether Nelarabine is effective in the treatment of patients with T-ALL/NHL in order to achieve a complete remission followed by an early stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* T-ALL; T-NHL
* age >= 18 years
* cytological treatment failure / relapse
* molecular treatment failure / relapse
* no promising therapy alternatives with approved medication available
* no CNS-manifestation, requiring intrathecal therapy or CNS-radiation
* no convulsive disease or neurotoxicity > grade III in patients history
* written informed consent
* no cytostatic therapy in the last 10 days
* no pregnancy or breastfeeding
* effective contraception
* recovery of toxicities of previous chemotherapy - except leukemia- related changes like bone marrow suppression or pathological transaminases in liver manifestation

Exclusion Criteria:

* Severe psychiatric illness
* uncontrolled or severe cardiac disease or infection
* active secondary neoplasms - except skin cancer (no melanoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Tolerability and Efficacy of Compound GW506U78 in relapsed/refractory T-ALL/NHL | after 1 cycle and 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD, PhD, Study Chair — University Hospital of Frankfurt, Medical Dept. II
Locations (11):
- Germany (11):
  - Robert Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität Regensburg, Regensburg, Bavaria
  - University Hospital of Frankfurt, Medical Dept. II, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinik Münster, Münster, North Rhine-Westphalia
  - Universitätsklinik Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Kiel, Kiel, Schleswig-Holstein
  - Klinikum der FSU Jena, Jena, Thuringia
  - HELIOS Klinikum Berlin-Buch, Berlin

REFERENCES:
- [Result] Gokbuget N, Basara N, Baurmann H, Beck J, Bruggemann M, Diedrich H, Guldenzoph B, Hartung G, Horst HA, Huttmann A, Kobbe G, Naumann R, Ratei R, Reichle A, Serve H, Stelljes M, Viardot A, Wattad M, Hoelzer D. High single-drug activity of nelarabine in relapsed T-lymphoblastic leukemia/lymphoma offers curative option with subsequent stem cell transplantation. Blood. 2011 Sep 29;118(13):3504-11. doi: 10.1182/blood-2011-01-329441. Epub 2011 Jun 28. PMID 21715318